CLINICAL TRIAL: NCT05540665
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Evaluating the Efficacy and Safety of Daxdilimab in Adult Participants With Active Proliferative Lupus Nephritis
Brief Title: Study of Daxdilimab (HZN-7734) in Participants With Active Proliferative Lupus Nephritis (LN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZNP-DAX-203; 2022-001377-31 (EudraCT Number)
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Daxdilimab Arm 1 (Experimental): Daxdilimab injections over a total of 104 weeks
  Interventions: Drug: Daxdilimab
- Daxdilimab Arm 2 (Experimental): Daxdilimab injections over a total of 104 weeks
  Interventions: Drug: Daxdilimab
- Placebo (Placebo Comparator): Placebo injections over a total of 104 weeks
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Drug: Daxdilimab — Daxdilimab will be administered subcutaneously as two injections for each dose.
  Other Names: HZN-7734
  Arms: Daxdilimab Arm 1
Drug: Daxdilimab — Daxdilimab will be administered subcutaneously as two injections for each dose.
  Other Names: HZN-7734
  Arms: Daxdilimab Arm 2
Drug: Placebo (Normal Saline) — Placebo will be administered subcutaneously as two injections for each dose.
  Arms: Placebo

SUMMARY:
Phase 2, multicenter, double-blind, randomized, placebo-controlled, parallel-group trial to evaluate the efficacy and safety of daxdilimab in patients with active, proliferative lupus nephritis (LN).

DETAILED DESCRIPTION:
Approximately 210 participants will be randomized to receive daxdilimab or placebo administered subcutaneously through Week 52 in addition to their standard of care background therapy (mycophenolate mofetil (MMF) and corticosteroids). At Week 64, all participants will be assigned to a quarterly dosing maintenance regimen of either daxdilimab or placebo based upon pre-defined renal response observed by Week 52. The maximum trial duration per participant is approximately 116 weeks including a 4-week screening period, the 104 weeks for the treatment period where participants will receive daxdilimab or placebo, and approximately 8 weeks for the follow-up period. Safety evaluations will be performed regularly throughout the course of the study.

Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and provide written informed consent
* Adult men or women 18 to 80 years of age
* Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial
* Fulfill the 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus (SLE)
* Have at least one of the following at Screening per central lab:

  * Antinuclear antibodies (ANA) ≥ 1:80
  * Anti-dsDNA antibodies elevated to above normal range as established by the central laboratory (ie, positive results)
  * Anti-Smith antibodies elevated to above normal (ie, positive results).
* Diagnosis of proliferative LN based on a renal biopsy obtained within 6 months prior to signing the informed consent form (ICF) or during the Screening Period:

  * Class III (± class V) or class IV (± class V) LN according to the World Health Organization (WHO) or 2003 International Society of Nephrology (ISN)/Renal Pathology Society (RPS) classification (based on local evaluation of renal biopsy).
* Urine protein to creatinine ratio ≥113.17 mg/mmol, obtained via a 24-hour urine collection at Screening.
* Estimated glomerular filtration rate ≥35 mL/min/1.73 m2
* Negative serum beta-human chorionic gonadotropin test at Screening (females of childbearing potential only).

Key Exclusion Criteria:

* History of allergy, hypersensitivity reaction, or anaphylaxis to any component of the investigational product or to a previous monoclonal antibody or human immunoglobulin therapy.
* Known intolerance to ≤1.0 gm/day of MMF or equivalent dose of mycophenolic acid (MPA).
* A diagnosis of pure Class V membranous LN based on a renal biopsy obtained within 6 months prior to signing ICF or during the Screening Period.
* History of dialysis within 12 months prior to signing the ICF or expected need for renal replacement therapy (dialysis or renal transplant) within a 12-month period after enrollment.
* History of, or current renal diseases (other than LN) that in the opinion of the Investigator could interfere with the LN assessment and confound the disease activity assessment (eg, diabetic nephropathy).
* Known history of a primary immunodeficiency or an underlying condition such as known human immunodeficiency virus (HIV) infection, a positive result for HIV infection per central laboratory, splenectomy, or any underlying condition that in the opinion of the Investigator significantly predisposes the participant to infection.
* Hepatitis B, Hepatitis C, active tuberculosis (TB), any severe herpes infection, clinically active infection, or opportunistic infection.
* Clinically significant cardiac disease including unstable angina, myocardial infarction, congestive heart failure within 6 months prior to Randomization.
* History of cancer within the past 5 years, except in situ carcinoma of the cervix, cutaneous basal cell or squamous cell carcinoma with curative therapy.
* Receipt of a live vaccine within 4 weeks prior to Day 1.
* The use of immunosuppressants, biologics, and DMARDS within the protocol defined washout periods.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (52):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Kidney Specialists, San Dimas, California
  - SUNY Upstate Medical University, Syracuse, New York
  - DaVita Clinical Research - El Paso, El Paso, Texas
  - Care and Cure Clinic, Houston, Texas
- Argentina (8):
  - Framingham Centro Médico, La Plata, Buenos Aires
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario, Santa Fe Province
  - DOM Centro de Reumatologia, Buenos Aires
  - Aprillus Asistencia e Investigacion de Arcis Salud SRL, Buenos Aires
  - Consultorios Médicos Dr. Doreski, Buenos Aires
  - Swiss Medical Center Barrio Parque, Ciudad Autónoma Buenos Aires
  - Centro de Investigaciones Médicas Tucumán, San Miguel de Tucumán
  - Clinica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán
- Brazil (11):
  - SER - Serviços Especializados em Reumatologia da Bahia S/S - ME, Salvador, Estado de Bahia
  - Clinica Senhor Do Bonfim CSB, Salvador, Estado de Bahia
  - Santa Casa de Misericórdia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
  - Oncovida- Centro de Onco-Hematologia de Mato Grosso, Cuiabá
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP - PPDS, Ribeirão Preto
  - Praxis Pesquisa Medica, Santo André
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Praxis Pesquisa Medica, São Paulo
- Clinical Hospital Centre Osijek, Osijek, Croatia
- Israel (3):
  - Lady Davis Carmel Medical Center, Haifa, Central District
  - Meir Medical Center, Kfar Saba, Central District
  - Sheba Medical Center - PPDS, Ramat Gan, Tel Aviv
- Malaysia (3):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Serdang, Kajang
  - Hospital Putrajaya, Putrajaya
- Philippines (3):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - St. Paul's Hospital, Iloilo City, Iloilo
  - GreenCity Medical Center, San Fernando City, Pampanga
- Poland (3):
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz, Lódzkie
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Warsaw
- Serbia (6):
  - University Clinical Center of Serbia - PPDS, Belgrade, Beograd
  - Institute of Rheumatology Belgrade - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - General Hospital Krusevac, Kruševac
  - University Clinical Center Nis, Niš
  - Clinical Centre of Vojvodina, Novi Sad
- Spain (4):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Manises, Valencia
- China Medical University Hospital, Taichung, Taiwan
- Thailand (4):
  - Rajavithi Hospital, Din Daeng, Krung Thep Maha Nakhon-Bangkok
  - Ramathibodi Hospital Mahidol University, Din Daeng, Krung Thep Maha Nakhon-Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Chiang Mai University, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with active proliferative lupus nephritis were recruited from centers in Argentina, Brazil, Malaysia, the Philippines, Poland, Serbia, and Thailand between April 2023 and January 2024, when the study was terminated.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to receive either daxdilimab 300 mg or 100 mg subcutaneously (SC) or placebo SC in addition to standard of care (SOC) background therapy for a Treatment Period of about 104 weeks. Participants were followed up for 12 weeks following last dose of investigational product (IP).
Groups:
- Placebo: Participants were randomized to receive placebo SC in addition to SOC background therapy at Day 1, Week 2, and Week 4. Thereafter, placebo was administered every 4 weeks (Q4W) through Week 52. At Week 64, dosing would have been adjusted based on renal response criteria: participants who achieved either partial renal response (PRR) or complete renal response (CRR) at both Weeks 48 and 52 would have continued to receive placebo at Week 64 and every 12 weeks (Q12W) through Week 104 (last dose at Week 100), in addition to SOC therapy. Participants who didn't achieve PRR or CRR at either Week 48 or 52 would have received daxdilimab 300 mg at Week 64 and then Q12W through Week 104 (last dose at Week 100), in addition to SOC therapy. However, the study was terminated prior to any participants reaching Week 64.
- Daxdilimab 100 mg: Participants were randomized to receive daxdilimab 100 mg SC in addition to SOC background therapy at Day 1, Week 2, and Week 4. From Week 8 through Week 52, daxdilimab was administered Q4W. At Week 64, dosing would have been adjusted based on renal response criteria: participants who achieved PRR or CRR at both Weeks 48 and 52 would have continued to receive daxdilimab 100 mg at Week 64 and Q12W through Week 104 (last dose at Week 100), in addition to SOC therapy. Participants who didn't achieve PRR or CRR at Week 48 or 52 would have received daxdilimab 300 mg at Week 64 and Q12W through Week 104 (last dose at Week 100), in addition to SOC therapy. However, the study was terminated prior to any participants reaching Week 64.
- Daxdilimab 300 mg: Participants were randomized to receive daxdilimab 300 mg SC in addition to SOC background therapy at Day 1, Week 2, and Week 4. From Week 8 through Week 52, daxdilimab was administered Q4W. At Week 64, dosing would have been adjusted based on renal response criteria: participants who achieved PRR or CRR at both Weeks 48 and 52 would have continued to receive daxdilimab 300 mg at Week 64 and Q12W through Week 104 (last dose at Week 100), in addition to SOC therapy. Participants who didn't achieve PRR or CRR at Week 48 or 52 would have received daxdilimab 300 mg at Week 64 and Q12W through Week 104 (last dose at Week 100), in addition to SOC therapy. However, the study was terminated prior to any participants reaching Week 64.
Period: Overall Study
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Started | 6 | 6 | 7
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 7
Not completed — Study terminated by sponsor | 6 | 6 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received any dose of IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg | Total
Number analyzed (Participants) | 6 | 6 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (5.91) | 31.5 (10.97) | 30.3 (6.47) | 32.8 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 17
  Male | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 4 | 2 | 7
  White | 5 | 2 | 5 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 6
  Not Hispanic or Latino | 3 | 6 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved CRR at Week 48 Through Week 52
Description: CRR was defined as meeting all of the following:
  * Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m^2 or no worse than 15% below Baseline
  * 24-hour urine protein to creatinine ratio (UPCR) ≤ 0.5 mg/mg
  * No discontinuation of trial intervention or use of restricted medication beyond the protocol-allowed threshold before assessment
Time Frame: Week 48 to Week 52
Population: Due to early termination data were not collected.
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Who Achieved Overall Renal Response (ORR) at Week 48 Through Week 52
Description: CRR was defined as meeting all of the following:
  * EGFR ≥ 60 mL/min/1.73 m^2 or no worse than 15% below Baseline
  * 24-hour UPCR ≤ 0.5 mg/mg
  * No discontinuation of trial intervention or use of restricted medication beyond the protocol-allowed threshold before assessment
  Partial renal response (PRR) was defined as meeting all of the following:
  * EGFR ≥ 60 mL/min/1.73 m^2 or no worse than 15% below Baseline
  * Improvement in 24-hour UPCR:
    * For participants with a Baseline UPCR ≤ 3.0 mg/mg: < 1.0 mg/mg
    * For participants with a Baseline UPCR > 3.0 mg/mg: > 50% improvement from baseline and ≤ 3.0 mg/mg
  * No discontinuation of trial intervention or use of restricted medication beyond the protocol-allowed threshold before assessment
Time Frame: Week 48 to Week 52
Population: Due to early termination data were not collected.
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in eGFR at Week 52
Description: Change over time in the levels of eGRF present in the blood.
Time Frame: Baseline and Week 52
Population: Due to early termination data were not collected.
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Proportion of Participants Achieving a Decrease in Daily Oral Corticosteroid (OCS) Dose of ≤ 2.5 mg Prednisone-Equivalent by Week 24 Maintained Through Week 52
Description: Sustained reduction of OCS dose:
  * Prednisone-equivalent dose ≤ 2.5 mg/day by Week 24 and not exceeding this dose through Week 52 and
  * No discontinuation of trial intervention or use of restricted medication beyond the protocol-allowed threshold before assessment
Time Frame: Week 24 to Week 52
Population: Due to early termination data were not collected.
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Serum Concentration of Daxdilimab
Description: Levels of daxdilimab present in the blood serum at different time points.
Time Frame: Week 0 pre-dose, and 6 hours post-dose; Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, and Week 36
Population: Pharmacokinetic (PK) Analysis Set: all participants who received any dose of daxdilimab and had at least 1 quantifiable PK observation following the initial dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 6 | 7
ng/mL
  Week 0 pre-dose | 7.80 (0.00) | 7.80 (0.00)
  Week 0 post-dose | 689.07 (498.40) | 3854.29 (3312.12)
  Week 2 | 4996.67 (1732.21) | 17610.00 (10382.53)
  Week 4 | 8531.67 (3993.99) | 22171.43 (9187.26)
  Week 8 | 3533.33 (1727.54) | 10330.00 (4167.07)
  Week 12: number analyzed (Participants) | 5 | 6
  Week 12 | 2988.00 (1223.83) | 10201.67 (4619.64)
  Week 16: number analyzed (Participants) | 3 | 2
  Week 16 | 1080.33 (1020.32) | 5051.50 (6644.68)
  Week 20: number analyzed (Participants) | 3 | 6
  Week 20 | 240.83 (184.66) | 2003.00 (3907.13)
  Week 24: number analyzed (Participants) | 2 | 1
  Week 24 | 93.85 (94.96) | 9660.00 (NA) — Standard deviation (SD) not calculated due to the low level of observations.
  Week 36: number analyzed (Participants) | 0 | 1
  Week 36 |  | 1040.00 (NA) — SD not calculated due to the low level of observations.

6. Secondary Outcome: Number of Participants With Detectable Anti-Drug Antibodies (ADA) Against Daxdilimab
Description: Assessed via blood test at multiple time points throughout the duration of the study.
Time Frame: Up to approximately 36 weeks
Population: Safety Analysis Set: All participants who received any dose of IP in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 6 | 6 | 7
Participants | 6 | 6 | 7

7. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical subject who was administered a pharmaceutical product, which may or may not have been causally related to the treatment. A serious AE (SAE) was any AE resulting in death, life-threatening situations, inpatient hospitalization or its prolongation, persistent/significant disability/incapacity, congenital abnormality/birth defect, or other significant medical events that may have jeopardized the participant or required medical/surgical intervention to prevent the outcomes listed above. Treatment-emergent AEs of special interest (AESI) included hypersensitivity reactions (e.g., anaphylaxis), severe viral infections/reactivations (Common Terminology for Adverse Events [CTCAE] Grade 3+), herpes zoster, opportunistic infections, and malignancies.
Time Frame: Up to approximately 36 weeks
Population: Safety Analysis Set: All participants who received any dose of IP in the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg
Number analyzed (Participants) | 6 | 6 | 7
Participants
  All TEAEs | 2 | 2 | 5
  All SAEs | 0 | 0 | 1
  All ≥ Grade 3 AESI | 0 | 0 | 0
  Fatal AEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 36 weeks
Description: All-cause mortality is reported for all participants randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of trial drug.
Groups:
- Daxdilimab Total: All participants who were exposed to daxdilimab.
- Total: Total
Arm/Group | Placebo | Daxdilimab 100 mg | Daxdilimab 300 mg | Daxdilimab Total | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/13 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/7 | 1/13 | 1/19
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 5/7 | 7/13 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Daxdilimab 100 mg (N=6) | Daxdilimab 300 mg (N=7) | Daxdilimab Total (N=13) | Total (N=19)
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Daxdilimab 100 mg (N=6) | Daxdilimab 300 mg (N=7) | Daxdilimab Total (N=13) | Total (N=19)
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Urinary sediment abnormal (Investigations) | 0 | 0 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early following a sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT05540665/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT05540665/SAP_001.pdf